CLINICAL TRIAL: NCT05551208
Title: A Prospective, Single-arm, Multicenter Phase Ⅱ Clinical Study of Fluzoparib Combined With Bevacizumab in Platinum-sensitive Recurrent Ovarian Cancer Patients Previously Treated With PARPi
Brief Title: Fluzoparib Combined With Bevacizumab in PSROC Previously Treated With PARPi
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Principal Investigator, Dongling Zou, Director of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0205
Record Dates: First submitted 2022-08-31; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Cancer
Keywords: PARP inhibitor; Fluzoparib; Bevacizumab; Platinum - sensitive recurrent EOC
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- maintenance treatment (Experimental): after 4-9 cycles chemotherapy containing platinum and bevacizumab, fluzopanib and bevacizumab were used for maintenance treatment
  Interventions: Drug: fluzopanib and bevacizumab

INTERVENTIONS:
Drug: fluzopanib and bevacizumab — fluzopanib and bevacizumab were used for maintenance treatment

SUMMARY:
There are more and more PARPi(PARP inhibitors) resistance for ovarian cancer patients after previous use of PARP inhibitors. Basic studies have found that there is synergistic effect of bevacizumab combined with PARPi. Therefore we designed the study to include 42 ovarian cancer patients who had PARPi for at least half a year and then relapsed (platinum-sensitive, previously 1-3 lines of chemotherapy). After getting complete remission or partial remission with chemotherapy containing platinum and bevacizumab, fluzopanib and bevacizumab were used for maintenance treatment. The progression-free survival, ORR, DCR, DoR, and safety were evaluated based on RECIST V1.1.

DETAILED DESCRIPTION:
Genetic testing of tissue samples before and after the maintenance therapy were also used to further explore the pattern of gene mutations and the subgroups who may benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Ovarian cancer patients with histopathological type: low/high grade serous carcinoma, endometrioid carcinoma,had received platinum-based regimens for at least 1-3 lines after primary cytoreductive surgery.
2. The patient had at least one measurable lesion according to the RECIST V1.1 criteria.
3. The time from the last cycle of chemotherapy to relapse/progression should be more than 6 months.
4. ECOG score 0~1,age 18~75 years old
5. The serum or urine pregnancy test must be negative within 7 days before enrollment for the women of childbearing age who should agree that contraception must be used during the trial
6. CBC Hb≥90g/L, ANC≥1.5×109/L, PLT≥100×109/L,
7. Serum ALT≤3×UL, AST≤3×ULN#Serum creatinine≤1.5×ULN#

Exclusion Criteria:

1. Had used bevacizumab within 6 months of enrollment
2. Has combined with other malignant tumor which diagnosed within 5 years and/or needed to be treated. The patients had untreated CNS metastases.
3. The patient had Recent intestinal obstruction, gastrointestinal perforation within 3 months, uncontrolled high blood pressure after medication (Systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg), Moderate to severe cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), moderate to severe deep vein thrombosis and moderate to severe pulmonary embolism occurred within 6 months before enrollment. Patient with coagulation dysfunction.
4. Myocardial infarction, severe arrhythmia and NYHA (New York heart association)≥2 for congestive heart failure
5. Activity or uncontrol severe infection

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 5 years
  progression-free survival was the maintenance time to progression or recurrence since the last platinum therapy based on RECIST v1.1

SECONDARY OUTCOMES:
OS | 5 years
  Overall survival
ORR | 5 years
  Objective Response Rate
DCR | 5 years
  Disease control rate
DoR | 5 years
  Duration of remission

OTHER OUTCOMES:
saftey | 5 years
  The severity of adverse events was determined according to CTCAE V5.0 criteria. During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, correlation with study treatment, duration, measures taken and outcome of the adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Zou Dongling, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Laar R, Zusterzeel PL, Van Gorp T, Buist MR, van Driel WJ, Gaarenstroom KN, Arts HJ, van Huisseling JC, Hermans RH, Pijnenborg JM, Schutter EM, Pelikan HM, Vollebergh JH, Engelen MJ, Inthout J, Kruitwagen RF, Massuger LF. Cytoreductive surgery followed by chemotherapy versus chemotherapy alone for recurrent platinum-sensitive epithelial ovarian cancer (SOCceR trial): a multicenter randomised controlled study. BMC Cancer. 2014 Jan 14;14:22. doi: 10.1186/1471-2407-14-22. PMID 24422892
- [Background] Harter P, Sehouli J, Vergote I, Ferron G, Reuss A, Meier W, Greggi S, Mosgaard BJ, Selle F, Guyon F, Pomel C, Lecuru F, Zang R, Avall-Lundqvist E, Kim JW, Ponce J, Raspagliesi F, Kristensen G, Classe JM, Hillemanns P, Jensen P, Hasenburg A, Ghaem-Maghami S, Mirza MR, Lund B, Reinthaller A, Santaballa A, Olaitan A, Hilpert F, du Bois A; DESKTOP III Investigators. Randomized Trial of Cytoreductive Surgery for Relapsed Ovarian Cancer. N Engl J Med. 2021 Dec 2;385(23):2123-2131. doi: 10.1056/NEJMoa2103294. PMID 34874631
- [Background] Coleman RL, Brady MF, Herzog TJ, Sabbatini P, Armstrong DK, Walker JL, Kim BG, Fujiwara K, Tewari KS, O'Malley DM, Davidson SA, Rubin SC, DiSilvestro P, Basen-Engquist K, Huang H, Chan JK, Spirtos NM, Ashfaq R, Mannel RS. Bevacizumab and paclitaxel-carboplatin chemotherapy and secondary cytoreduction in recurrent, platinum-sensitive ovarian cancer (NRG Oncology/Gynecologic Oncology Group study GOG-0213): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Jun;18(6):779-791. doi: 10.1016/S1470-2045(17)30279-6. Epub 2017 Apr 21. PMID 28438473
- [Background] Aghajanian C, Blank SV, Goff BA, Judson PL, Teneriello MG, Husain A, Sovak MA, Yi J, Nycum LR. OCEANS: a randomized, double-blind, placebo-controlled phase III trial of chemotherapy with or without bevacizumab in patients with platinum-sensitive recurrent epithelial ovarian, primary peritoneal, or fallopian tube cancer. J Clin Oncol. 2012 Jun 10;30(17):2039-45. doi: 10.1200/JCO.2012.42.0505. Epub 2012 Apr 23. PMID 22529265
- [Background] Alvarez Secord A, O'Malley DM, Sood AK, Westin SN, Liu JF. Rationale for combination PARP inhibitor and antiangiogenic treatment in advanced epithelial ovarian cancer: A review. Gynecol Oncol. 2021 Aug;162(2):482-495. doi: 10.1016/j.ygyno.2021.05.018. Epub 2021 Jun 3. PMID 34090705
- [Background] Ray-Coquard I, Pautier P, Pignata S, Perol D, Gonzalez-Martin A, Berger R, Fujiwara K, Vergote I, Colombo N, Maenpaa J, Selle F, Sehouli J, Lorusso D, Guerra Alia EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marme F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428. doi: 10.1056/NEJMoa1911361. PMID 31851799
- [Background] Fong PC, Boss DS, Yap TA, Tutt A, Wu P, Mergui-Roelvink M, Mortimer P, Swaisland H, Lau A, O'Connor MJ, Ashworth A, Carmichael J, Kaye SB, Schellens JH, de Bono JS. Inhibition of poly(ADP-ribose) polymerase in tumors from BRCA mutation carriers. N Engl J Med. 2009 Jul 9;361(2):123-34. doi: 10.1056/NEJMoa0900212. Epub 2009 Jun 24. PMID 19553641
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338